CLINICAL TRIAL: NCT02606396
Title: Palliation of Malignant Dysphagia With Spray Cryotherapy in Patients With Advanced Esophageal Cancer: A Pilot Study
Brief Title: Cryotherapy for Malignant Dysphagia in Patients With Advanced Esophageal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201510035
Record Dates: First submitted 2015-11-09; First posted 2015-11-17 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Esophageal Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — Cryotherapy; Endoscopy, Digestive System; Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Cryotherapy — Cryotherapy employs thermal ablation to treat esophageal cancer and BE. Ablation is achieved by intracellular disruption and ischemia that is produced by freeze-thaw cycles using liquid nitrogen or carbon dioxide
Procedure: Esophagogastroduodenoscopy (EGD) — EGD is a diagnostic procedure that allows the physician to diagnose and treat problems in the upper gastrointestinal (UGI) tract. The doctor uses a long, flexible, lighted tube called an endoscope.
Procedure: Endoscopic ultrasound (EUS) — EUS is a procedure that allows a doctor to obtain images and information about the digestive tract and the surrounding tissue and organs, including the lungs. Ultrasound testing uses sound waves to make a picture of internal organs.

SUMMARY:
Esophageal adenocarcinoma (EAC) is one of the few cancers with a rising incidence in the United States, with an estimated 17,000 new cases diagnosed in 2012. Most patients with esophageal cancer present with tumors which are not amenable to surgery and are treated with chemotherapy and radiation. The most common and bothersome symptoms from esophageal cancer is dysphagia (difficulty swallowing). Chemotherapy and radiation are effective in shrinking tumors and allowing patients with EAC to swallow more easily; however it usually takes 1-2 months for swallowing to improve with this treatment.

Another method of shrinking esophageal tumors and allowing for better swallowing is endoscopic spray cryotherapy (freezing the tumor from inside the esophagus with the aid of an endoscope); cryotherapy is a well established method for treating cancerous and pre-cancerous esophageal disease. This is a particularly attractive treatment option, as patients with esophageal cancer usually undergo endoscopy on several occasions before starting treatment in order to biopsy and evaluate the tumor.

The goal of this study is to evaluate the effectiveness of cryotherapy in treating EAC related dysphagia in patients who are getting ready to start chemotherapy and radiation.

In order to do this the investigators are planning to invite patients who are already undergoing endoscopy for pre-chemotherapy evaluation of known EAC. Patients would undergo cryotherapy after the diagnostic portion of the endoscopy has been completed. After the cryotherapy patients will be contacted by phone in order to evaluate change in symptoms, 2 and 4 weeks after cryotherapy.

DETAILED DESCRIPTION:
Endoscopic spray cryotherapy (EC) is a novel modality for destruction of tissue in the gastrointestinal tract. EC involves the endoscopic application of cryogen [liquid nitrogen (LN)], which destroys tissue by rapid freezing and slow thawing. Immediate effects from tissue freezing include failure of cellular metabolism, membrane damage and local ischemia. Delayed effects may include apoptosis of cancer cells and immune mediated tumor destruction. EC has been used for the treatment of mucosal EAC and palliation of malignant dysphagia since 2007 in multiple tertiary centers, including Washington University in St Louis, with positive results. EC is an attractive modality for the palliation of malignant dysphagia in EAC due to the fact that newly diagnosed patients undergo upper endoscopy (EGD) and endoscopic ultrasound (EUS) as part of initial staging; thus EC could be delivered at the time of the staging endoscopy, without burdening the patient with an additional procedure. However, prospective studies on the efficacy of EC in the short term palliation of malignant dysphagia in EAC have not been performed.

Thus, the goal of this pilot study is to evaluate the effectiveness of EC in the short term palliation of malignant dysphagia in patients with unresectable EAC.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age with malignant dysphagia due to locally advanced EAC (≥T3 and/or N1) who are undergoing upper endoscopic ultrasound or upper endoscopy for pre-treatment staging or symptom evaluation

Exclusion Criteria:

* Prior esophageal or gastro-esophageal junction surgery.
* Prior diagnosis of oropharyngeal dysphagia.
* Prior diagnosis of esophageal achalasia.
* Esophageal strictures unrelated to EAC
* Distant metastasis
* Dysphagia only to solid or semi-solid foods
* Need for esophageal dilation in order to pass the diagnostic upper endoscope distal to the tumor.
* Coagulopathy (INR>2, platelets < 50,000)
* Inability to provide informed consent.
* Marfan's syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change in dysphagia severity according to validated symptom score | 2 weeks after cryoablation session

SECONDARY OUTCOMES:
Ability to maintain oral intake evaluated by a member of the study team utilizing dysphagia assessment and oral intake assessment instruments who will contact each patient at 1-month intervals while the patient receives chemoradiation | Up to 12 weeks
Assessment of pathologic complete response and clinical complete response at the completion of neo-adjuvant chemoradiation number one. | Up to 24 weeks
  Results of the re-staging PET-CT will be abstracted from the medical record to document presence or absence of a pathologic complete response
Assessment of pathologic complete response and clinical complete response at the completion of neo-adjuvant chemoradiation number two. | Up to 24 weeks
  Results of the surgical explant will be abstracted from the medical record to document presence or absence of a pathologic complete response.
Incidence of procedure related adverse events, classified according to the American Society of Gastrointestinal Endoscopy lexicon | 1 week after each procedure; 2 to 3 weeks after each procedure and 8 weeks after completion of the last cryoablation session

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir M Kushnir, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Center for Advanced Medicine, St Louis, Missouri, United States